CLINICAL TRIAL: NCT00221793
Title: Study of Ponderal Load in Parkinsonian Patients After Deep Brain Stimulation of the Subthalamic Nucleus
Brief Title: Weight Changes in Parkinsonian Patients, Treated With Deep Brain Stimulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Jean-Pierre LEROY / Clinical Research and Innovation Director, University Hospital, Bordeaux
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 9212-02
Record Dates: First submitted 2005-09-13; First posted 2005-09-22 (Estimated); Last update posted 2008-09-18 (Estimated); Status verified 2008-09

CONDITIONS: Parkinson Disease
Keywords: Parkinson; deep subthalamic stimulation; pharmacological treatment
MeSH Terms: conditions — Parkinson Disease | interventions — Deep Brain Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Deep Brain Stimulation of the Subthalamic Nucleus
  Interventions: Procedure: Deep brain stimulation
- 2 (Active Comparator): Later Deep Brain Stimulation of the Subthalamic Nucleus
  Interventions: Procedure: Deep brain stimulation

INTERVENTIONS:
Procedure: Deep brain stimulation — Brain Stimulation of the Subthalamic Nucleus

SUMMARY:
The aim of this trial is to verify that neurostimulated parkinsonian patients gain weight and to study its link with an energetic balance change.

DETAILED DESCRIPTION:
The aim of this trial is to verify that neurostimulated parkinsonian patients gain weight and to study its link with an energetic balance change.

Twenty parkinsonian patients will be randomised : the delay between inclusion and neurostimulation wil be lengthened 3 months for one group, compared to the second one. The energy expenditure, at rest and after ingestion of a test meal, will be compared between the group of patients that had been neurostimulated and the group whose intervention has been postponed. Weight changes, energy intake, leptin level, neurophysiological parameters will be compared between both groups, and the nature and repartition of the weight gain will be assessed in the neurostimulated group. An eventual link between motor factors, pharmacological factors, and gain weight will be studied.

ELIGIBILITY:
Inclusion Criteria:

* Age between 35 and 70; male or female; parkinson disease, with levo dopa response (at least 30%); severe but stable incapacity; no dementia, no psychosis, no depression; normal brain scanner done during the last 2 years.

Exclusion Criteria:

* diabetes thyroid disease pacemaker coagulation troubles previous drug abuse

Ages: 35 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2002-12; Primary Completion 2006-12 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Measurement of energy expenditure with indirect calorimetry in open chamber: at rest in the morning, without 24h-dopaminergic treatment, and after dopaminergic treatment intake; and post prandial thermogenesis after a test meal. | After surgery and at 3 months

SECONDARY OUTCOMES:
Weight gain | At visit 1 and at 3 months
increase of energy intake | At visit 1 and at 3 months
leptin, glucose, insulin blood levels | At visite 1 and at 3 months
cognitive and psychological assessments | before surgery and after 3 months
UDPRS scale | before surgery and after 3 months

CONTACTS AND LOCATIONS:
Overall Officials: François TISON, Pr, Principal Investigator — Service de neurologie Hôpital Haut-Lévêque Pessac; Jacques DEMOTES-MAINARD, Pr, Study Chair — CIC Inserm-CHU de Bordeaux Pessac
Locations (1):
- Service de neurologie Hôpital Haut-Lévêque, Pessac, France